CLINICAL TRIAL: NCT05779319
Title: The 1000 Eyes Lens Power Trial: Introducing Artificial Intelligence to Intraocular Lens Power Calculation
Brief Title: 1000 Eyes Lens Biometry Study: Artificial Intelligence for Intraocular Lens Power Calculation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Mein Hanusch-Krankenhaus (Other); Medical University of Graz (Other); Landesklinikum Sankt Polten (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Opthalmology-013
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Cataract
Keywords: lens power calculation; biometry; artificial inteligence
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: non contact measurement with the IOL Master 700 — postoerpative we will perform non contact measurement with the IOL Master 700

SUMMARY:
The main purpose of the study is to develop an AI approach to improve intraocular lens power calculations.

DETAILED DESCRIPTION:
Cataract surgery is one of the most commonly performed surgeries worldwide and has a high postoperative patient satisfaction rate. Despite significant improvement in measurement methods and artificial lens power calculation formulas, miscalculations and subsequently refractive error still occur after cataract surgery.

Most current artificial lens calculation methods use regression formulas. The concept of artificial intelligence (AI) has only recently found use and only in a rudimentary way. Examples include the Hill-RBF calculator and the Ladas superformula, but at least the "superformula" does not use a true AI approach and the results are no better than those obtained with conventional methods.

The main purpose of the study is to develop an AI approach to improve intraocular lens power calculations. The data will be used for the following analysis:

* To compare the new AI method with conventional and modern formula (main question)
* To compare the refractive error for different eye lengths
* To use a ray tracing method to quantify sources of error in patients with a refractive surprise of at least 1.0 diopter
* To evaluate a novel concept of outlier testing using a modified nonparametric Walsh test

This study will be multi-center and partially prospective. Data from 1000 patients who have already had cataract surgery will be analyzed.

All patients will be invited for a visit to the recruitment clinic and the measurements will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic (at least one eye): cataract surgery between 4 weeks and 24 months prior to recruitment
* If both eyes would be suitable for the study only the right eye will be included, if only one eye is suitable for the study, this eye will be included
* Pre-operative swept-source OCT biometry available (no ultrasound measurement for axial eye length)
* Uncomplicated cataract surgery
* Age 21 years and older

Exclusion Criteria:

* Multifocal IOLs
* Combined surgery (cataract plus glaucoma/vitreoretinal/corneal surgery)
* Best corrected distance visual acuity below 0.5 Snellen
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will routinely undergo cataract surgery at one of the participating centers will be asked during the preliminary examination if they want to participate in the study. If they meet the inclusion criteria, they will be called to the clinic for a postoperative measurement within 4 weeks to 24 months after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
a new artificial intelligence based approach for intraocular lens power calculation | 2 years
  Developing an artificial intelligence algorithm to predict post-operative refraction

CONTACTS AND LOCATIONS:
Overall Officials: Nino Hirnschall, MD, Principal Investigator — JKU Linz
Locations (1):
- Kepler University Klinik Departement of Opthalmology, Linz, Upperaustria, Austria